CLINICAL TRIAL: NCT02212262
Title: Role of Osteocytes in Myeloma Bone Disease
Status: Completed | Type: Observational
Sponsor: Attaya Suvannasankha (Other)
Responsible Party: Sponsor-Investigator, Attaya Suvannasankha, Assistant Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: IUCRO-0498
Record Dates: First submitted 2014-07-31; First posted 2014-08-08 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multiple Myeloma Patients: Patients with multiple myeloma will undergo a blood draw and a bone marrow aspirate. Extra bone marrow will be taken for study purposes only.
- Healthy subjects: Healthy subjects and multiple myeloma patients will undergo a blood draw

SUMMARY:
Progress in the treatment of myeloma and myeloma bone disease has substantially increased overall survival, but relapse is inevitable and better treatment is needed. The bone microenvironment is tremendously complex, so that targeting single interactions between tumor and bone is unlikely to be effective. Treatments need to block centrally important, multifunctional pathways. The investigators data point to a central role of the osteocyte to induce heparanase, a multifunctional mediator of myeloma bone disease. Increased heparanase due to FGF23 may make systemic inhibitors of heparanase less effective in bone than elsewhere. FGF23 neutralizing antibodies have been developed for non-cancer conditions of FGF23 excess, such as chronic kidney disease (Shimada & Fukamoto, 2012), and could be used in MM alone or in combination with heparanase inhibitors. Complete neutralization of FGF23 has adverse effects, but neutralization of FGF23 excess may be practical, or in the future, suppression of excess FGF23 biosynthesis by osteocytes.

The investigators hope to determine serum FGF23 and heparanase, Dkk1 and plasma klotho levels in patients with newly diagnosed and relapsed myeloma compared to healthy controls with this exploratory study.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years but ≤ 95 years at the time of consent
2. Subjects must be English-speaking
3. Must voluntarily sign the most current informed consent and HIPAA documents prior to study participation.
4. Have no prior history of malignancy in the past 5 years with the exception of basal cell and squamous cell carcinoma of the skin. Other cancers with low potential for metastasis, such as in situ cancers can also be enrolled as healthy volunteers.
5. Have no known liver or kidney disorders

Exclusion Criteria:

1. Pregnant females will be excluded from the study.
2. Subjects allergic to xylocaine will be excluded.
3. Subjects with an acute illness (Ex. upper respiratory infection, viral illness) in the past seven days will be excluded.
4. History of bleeding disorders.
5. Subjects deemed incompetent by treating physician
6. Institutionalized, mentally disabled subjects
7. Subjects who are prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oncology Clinics at Indiana University Roudebuch VA Medical Center Community sample
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-05 (Actual)

PRIMARY OUTCOMES:
Molecular interactions between multiple myeloma and osteocytes | Up to 4 years
  To determine FGF23 and heparanase, Dkk1 and plasma klotho levels increase in patients with newly diagnosed and relapsed myeloma compared to healthy controls.

SECONDARY OUTCOMES:
Multiple Myeloma osteocytes and tumor staging | Up to 4 years
  To correlate the FGF23, heparanase, Dkk1 and plasma klotho to tumor staging
Multiple Myeloma osteocytes and Type I collagen fragments on bone resorption | Up to 4 years
  To correlate the FGF23, heparanase, Dkk1 and plasma klotho to extent of bone resorption using serum type I collagen fragments ICTP and CTX

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, M.D., Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - VA Roudebush Medical Center, Indianapolis, Indiana